CLINICAL TRIAL: NCT05573841
Title: Transfusion for Major Haemorrhage in Trauma - Characteristics and Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Hedberg, Principal Investigator, MD, PhD, Karolinska University Hospital
Other Study IDs: K 2022-5528
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Trauma; Hemorrhage; Shock, Traumatic; Acute Coagulopathy
MeSH Terms: conditions — Wounds and Injuries; Hemorrhage; Shock, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Trauma is the leading cause of death in young adults worldwide and the most common causes of mortality are haemorrhage and brain injury. About 40% of trauma related deaths are due to massive haemorrhage and approximately 30% of trauma patients have an associated trauma induced coagulopathy. In order to improve outcome, the optimal care for the bleeding patient need to be further understood.

Aim: The overall aim of this project is to evaluate characteristics and outcomes in patients receiving blood transfusion in the early phase after major trauma at a Level 1 trauma center in Sweden.

The specific aims are:

i) To describe outcome, characteristics and effects on the coagulation system in patients receiving early blood transfusion compared to those not receiving transfusion in the early phase.

ii) To describe outcome, characteristics and effects on the coagulation system in patients receiving prehospital blood transfusion compared to patients where transfusion is initiated in the trauma unit.

iii) To describe the effect from concurrent treatment with procoagulant drugs and intravenous fluids on outcome, characteristics and effects on the coagulation system in patients receiving blood transfusion after major trauma.

Method: This is an observational study of trauma patients admitted to the Trauma Unit at the Karolinska University Hospital Solna, Stockholm, Sweden. Data from patients receiving blood transfusion (erythrocytes, plasma or whole blood) in the early phase of the resuscitation will be collected. All patients receiving transfusion within two hours from arrival will be included. Data on trauma details, injuries, physiological parameters, coagulations tests and treatment will be collected prospectively and from existing registries. The control group will consist of patients not receiving transfusion during the first two hours of care.

ELIGIBILITY:
Inclusion Criteria:

* All trauma patients admitted to the trauma unit at the Karolinska University Hospital Solna.

Exclusion Criteria:

* Patients with injuries från hanging, drowning, burns or smoke inhalation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All trauma patients admitted to the trauma unit at the Karolinska University Hospital Solna will be studied. Patients receiving unmatched blood (erythrocytes, plasma or whole blood) either in the prehospital phase or during the first two hours of hospital care will be compared to patients not receiving blood products.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Survival | 30 day

SECONDARY OUTCOMES:
Trauma-induced coagulopathy defined as INR > 1.2 | Admission to 24 hours
Survival | 24 hour
Volume of transfusion | Admission to 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No